CLINICAL TRIAL: NCT07220655
Title: Cognition and Ultrasound
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PSYCH-2024-33067
Record Dates: First submitted 2025-10-22; First posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Low-Intensity Focused Ultrasound (Experimental)
  Interventions: Device: Low-Intensity Focused Ultrasound (FUS or LIFU)

INTERVENTIONS:
Device: Low-Intensity Focused Ultrasound (FUS or LIFU) — We will use an established, currently-marketed device to deliver LIFU neuromodulation.

SUMMARY:
Our primary goal is to investigate the role of Low-Intensity Focused Ultrasound (LIFU) neuromodulation on deep brain targets, and its potential to improve cognition

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Speak English (as assessed by their ability to read/answer survey questions)
* May be required to score in the appropriate range on self-report measures

Exclusion Criteria:

* They have a neurological disorder which may impact their fMRI scan or cause their reaction to LIFU to differ from that of healthy adults.
* They take any psychoactive medication.
* They are unable to undergo fMRI scanning due to a contraindication such as claustrophobia, unremovable piercings, pregnancy, the presence of medical devices such as pacemakers, or a movement or sleep disorder.
* Are pregnant, or may have reason to believe that they are pregnant.
* They have a diagnosis of a psychiatric condition other than depression or anxiety

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Deep Brain Targets Reached | Hour 1
  MRI-based readouts testing whether LIFU neuromodulation can successfully engage targets in deep brain
Multi-Source Interference Test (MSIT) Performance | Hour 1
  Behavioral readouts of successful LIFU neuromodulation of our target regions
28/Posit Science Performance | Hour 1
  Behavioral readouts of successful LIFU neuromodulation of our target regions

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bronstein, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No